CLINICAL TRIAL: NCT04034394
Title: Electromoxibustion and Knee Health Education for Knee Osteoarthritis in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Emoxi Knee OA
Record Dates: First submitted 2019-07-18; First posted 2019-07-26 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromoxibustion (Experimental): Participants in this group will receive electromoxibustion using a knee-brace-like device which produces thermal stimulation with a moxa pad inside (Fort Mayer, Guangzhou, China).
  Interventions: Other: Electromoxibustion
- Knee health education (Active Comparator): Participants in this group will attend 2 sessions (120 minutes each, 1-week apart) of health education related to knee OA symptom management.
  Interventions: Other: Knee health education

INTERVENTIONS:
Other: Electromoxibustion — Electromoxibustion is a electric device that mimic the burning or moxa. Subjects in this group will receive electromoxibustion using a knee-brace-like device which produces thermal stimulation with a moxa pad inside. The treatment will be delivered 3 times per week for 4 weeks.
  Arms: Electromoxibustion
Other: Knee health education — Subjects in this group will attend 2 lessons (120 minutes each) of health education related to knee OA symptom management in a small group of 5-7 subject. The course content is developed from the course materials from the websites of Elderly Health Service, Department of Health, Hong Kong SAR.
  Arms: Knee health education

SUMMARY:
This is a randomized controlled trial comparing the short-term effect of electromoxibustion and knee health education for relieving knee pain in older adults with knee osteoarthritis.

DETAILED DESCRIPTION:
Objective: This pilot randomized controlled trial (RCT) will preliminary examine the effects of an electromoxibustion device and knee health education on reliving knee osteoarthritis (OA) pain.

Method Design: This pilot RCT will embed a two-arm randomized control trial. The project will recruit 48 participants with knee OA. Eligible participants will be randomized into 2 groups - (1) Electromoxibustion, or (2) knee health education at 1:1 ratio.

Interventions: Participants in the electromoxibustion group will receive electromoxibustion using a knee-brace-like device which produces thermal stimulation with a moxa pad inside (Fort Mayer, Guangzhou, China); participants in the Knee health education group will attend 2 sessions (120 minutes each, 1-week apart) of health education related to knee OA symptom management.

Outcome measures: (1) Pain severity numerical rating scale (NRS) (Primary outcome); (2) Western Ontario and McMaster University Osteoarthritis Index (WOMAC) for pain, physical function, and stiffness related to knee osteoarthritis; (3) Short Form-6 Dimensions for quality of life; (4) Timed Up & Go Test (TUG); (5) Fast Gait Speed (FGS) for knee functioning.

Statistical Analysis of quantitative data: Descriptive statistics will be used to describe the socio-demographic characteristics of the participants. A mixed-effects model with consideration of repeated measures and dropout by including all available data points (intention-to-treat analysis) to compare the electromoxibustion with the knee health education control group. SPSS version 23.0 will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. ethnic Chinese;
2. aged 60 years or above;
3. ability to comprehend Chinese;
4. fulfilling any 3 of the following criteria: i. morning stiffness </= 30 min; ii. crepitus on active joint motion; iii. bone tenderness; iv. bone enlargement; or v. no palpable joint warmth (This classification yielded 84% sensitivity and 89% specificity for OA knee diagnosis (Altman et al., 1986);
5. having knee pain for at least 3 months;
6. Knee pain ≥4 on a Likert pain scale from 1-10; and
7. willing to provide informed consent.

Exclusion Criteria:

1. medical diagnoses or conditions that preclude individuals from active participation (e.g. dementia, post-stroke syndrome, alcohol or drug abuse);
2. knee pain related to other conditions (cancer, fracture, rheumatoid arthritis, rheumatism) as screened according to the red flags for further investigation or referral in the National Clinical Guideline Centre 2014 Guidelines for Osteoarthritis of the knee (National Clinical Guideline Centre, 2014);
3. presence of skin lesions or infections at the treatment sites;
4. ever had knee replacement surgery or knee joint implant; and
5. ever received moxibustion, electromoxibustion or steroid injection for knee pain over the past 6 months; Further investigation or referral, either at the screening or during the study, will be made when necessary.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Pain severity numerical rating scale, NRS | Week 4
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). It has been shown that a composite scoring system including best, worse, and current level of pain over the last 24 hours was sufficient to pick up changes in pain intensity with maximal reliability.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Week 4
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales.The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
Short Form-6D | Week 4
  The SF-6D, which is derived from the 36-item Short Form Health Survey (SF-36), is one of the most widely used generic measures of HRQoL in clinical trials. The score ranges from 0 to 1.
Timed Up & Go Test (TUG) | Week 4
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
Fast Gait Speed (FGS) | Week 4
  Subjects will be asked to walk 4 metres at their normal pace. Their gait speed in metres per second will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Wing Fai YEUNG, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Cheung T, Ho YS, Yuen CS, Lam CS, Chun-Lung So B, Chen SC, Leung DYP, Kwai-Ping Suen L, Tin-Yau So L, Chun-Hei Ho A, Yeung WF. Electromoxibustion for knee osteoarthritis in older adults: A pilot randomized controlled trial. Complement Ther Clin Pract. 2020 Nov;41:101254. doi: 10.1016/j.ctcp.2020.101254. Epub 2020 Nov 6. PMID 33190009